CLINICAL TRIAL: NCT00364650
Title: Probiotic Prophylaxis for Immunosuppressant Associated Diarrhea (IAD) Following Kidney Transplantation: a Single Center Randomized Controlled Trial
Brief Title: Probiotic Prophylaxis for Immunosuppressant Associated Diarrhea (IAD) Following Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish Medical Center (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: William H Marks MD PhD, Swedish Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEL346 (Main)
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Immunosuppressant Associated Diarrhea
Keywords: Renal transplantation; Diarrhea; Immunosuppression; Probiotics
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- I (Placebo Comparator): Placebo
  Interventions: Other: Placebo
- II (Experimental): Probiotic supplement
  Interventions: Drug: Probiotic Supplement

INTERVENTIONS:
Drug: Probiotic Supplement — 2 capsules twice daily
  Arms: II
Other: Placebo — placebo
  Arms: I

SUMMARY:
We hypothesize that the administration of a combination of high numbers of probiotic bacteria will maintain normal bowel function and significantly moderate or obviate Immunosuppression Associated Diarrhea following kidney transplantation.

DETAILED DESCRIPTION:
Immunosuppression following organ transplantation is associated with a myriad of gastrointestinal complications including severe diarrhea. Mycophenolate mofetil (MMF) is the immunosuppressant most often associated with this plaguing symptom. A retrospective study of patients from 10 US transplant centers receiving MMF immunosuppression after kidney transplantation showed that nearly 50% of patients suffered from at least one gastrointestinal symptom within the first 6 months after transplantation. (Tierce 2005) The majority of these patients have diarrhea. However, Immunosuppression Associated Diarrhea (IAD) is often observed in association with other immunosuppressive agents as well. It is the investigator's observation that IAD is equally problematic whether the immunosuppressive regimen includes MMF or not. When IAD is severe it can be difficult for the recipient to maintain adequate levels of immunosuppression. Not infrequently, IAD is so distressing that a recipient's immunosuppressive medications are tapered, changed or stopped. During these times of drug manipulation, patients are at risk for early acute rejection. Approximately 30% of renal transplant patients who have their MMF regimen adjusted or discontinued suffer an episode of acute rejection. Reversing a rejection episode is expensive and adds significant risks for the recipient and long-term allograft survival. Thus, a strategy to support and maintain normal healthy bowel function moderating or obviating IAD is highly desirable.

Repopulation of the normal intestinal microflora in kidney transplant patients after kidney transplantation may maintain normal bowel function. This study is designed to test the hypothesis that the administration of a food supplement probiotic consisting of high amounts of six strains of lactic acid bacteria normally found in the human colon will favorably support and maintain bowel function moderating or obviating IAD.

ELIGIBILITY:
Inclusion Criteria:

* all subjects aged >/= 18 years who qualify to receive a living (related or unrelated) or cadaveric kidney allograft using steroid free induction immunosuppression.
* single organ recipient (kidney only)
* subjects receiving first or second renal transplant
* women of child-bearing potential should have a negative serum pregnancy test within 1 week prior to beginning study medications
* subjects with no known contraindications to treatment with any of the study drugs
* subjects providing written consent
* subjects who are compliant and able to complete all the necessary assessment procedures

Exclusion Criteria:

* Subjects < 18 years of age
* Subjects who do not meet criteria for steroid free protocol
* subjects with known intolerance to lactobacillus
* subjects with history of chronic diarrhea
* subjects with history of gastrointestinal disorder that may interfere with their ability to absorb oral medication: inflammatory bowel disease, irritable bowel syndrome, short gut syndrome, or ileo jejunal surgery
* subjects with known laxative abuse
* subjects with pancreatic insufficiency
* subjects who are pregnant, lactating or nursing
* subjects with active peptic ulcer disease
* child bearing women not willing to use a reliable form of contraception
* subjects with prior history of C. difficile
* subjects receiving other medications considered to be experimental for control of diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To maintain normal bowel function and significantly moderate or obviate Immunosuppression Associated Diarrhea following kidney transplantation, utilizing a daily questionnaire, stool cultures and C. Difficile. | 5 months

SECONDARY OUTCOMES:
Determine the impact of IAD on therapeutic drug levels. Taper or change of immunosuppressive medications due to IAD. | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: William H Marks, MD, PhD, Principal Investigator — Swedish Medical Center
Locations (1):
- Swedish Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Cooper TE, Scholes-Robertson N, Craig JC, Hawley CM, Howell M, Johnson DW, Teixeira-Pinto A, Jaure A, Wong G. Synbiotics, prebiotics and probiotics for solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 20;9(9):CD014804. doi: 10.1002/14651858.CD014804.pub2. PMID 36126902